CLINICAL TRIAL: NCT05448625
Title: Safety and Efficacy of Sirolimus-eluting Biodegradable Abluminal Coating Stents in Patients With a High Risk of Ischemic Events: a Single-center, Prospective, Observational Trial (GENTLE Registry)
Brief Title: Genoss DES in Patients With a High Risk of Ischemic Events (GENTLE Registry)
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Collaborators: Severance Hospital (Other); Genoss Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Yongcheol Kim, Clinical Associate Professor, Yonsei University
Other Study IDs: 9-2022-0014
Record Dates: First submitted 2022-06-21; First posted 2022-07-07 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Drug-eluting Stent; Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- High Ischemic Group: 1. Acute myocardial infarction (AMI)
  2. ≥ 2 stents implanted
  3. bifurcation lesion
  4. Left main lesion
  5. Lesion treated with rotational atherectomy
  6. Chronic total occlusion (CTO) lesion
  Interventions: Device: Genoss DES

INTERVENTIONS:
Device: Genoss DES — The Genoss DES (Genoss, Korea) L-605 cobalt chromium (CoCr) platform with a strut thickness of 70 µm Sirolimus drug with concentration of 1.15µg/mm2 Abluminal biodegradable PLA and PLGA polymers.

SUMMARY:
This is a prospective cohort study to evaluate the long-term effect and safety of Genoss drug-eluting stents (DES) in patients with coronary artery disease with high ischemic features.

DETAILED DESCRIPTION:
It is known that ischemic events after percutaneous coronary intervention (PCI) or coronary artery bypass surgery (CABG) increase as the anatomical, physiological, or functional complexity of coronary artery disease increases. Recently, the concept of complex higher-risk and clinically indented procedure (CHIP) has been proposed, which includes patients with various medical conditions, patients with various heart conditions, and patients with technically complex PCI. Until now, Genoss stents have no data on the evaluation of stents in patients with coronary artery disease and high ischemic features.

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥ 19 years
* Subject has signed informed consent for data release

Exclusion Criteria:

* Subject did not sign informed consent for data release
* Known intolerance to aspirin, clopidogrel, ticlopidine, heparin or any other anticoagulation / antiplatelet therapy required for PCI, cobalt chromium, Sirolimus or contrast media
* Pregnancy
* Subject with life expectancy less than 12 months
* Subject with cardiogenic shock

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All-comers patient population with all subjects requiring coronary revascularization with a Drug Eluting Stent (DES)
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2022-05-26 (Actual); Primary Completion 2025-05-14 (Actual); Study Completion 2025-09-23 (Actual)

PRIMARY OUTCOMES:
Number of participants with device-oriented compopsite endpoint (TLF) | 12 months
  A composite rate of cardiac death (CD), target-vessel myocardial infarction (TV-MI), Ischemic driven target lesion revascularization (ID-TLR)

SECONDARY OUTCOMES:
Number of participants with patient-oriented composite endpoint | 12 months
  A composite rate of all death, all myocardial infarction, and all revascularization
Number of participants with all death | 12 months
  A composite rate of all death
Number of participants with cardiac death | 12 months
  A composite rate of cardiac death
Number of participants with non-cardiac death | 12 months
  A composite rate of non-cardiac death
Number of participants with all myocardial infarction | 12 months
  A composite rate of all myocardial infarction
Number of participants with target-vessel myocardial infarction (TV-MI) | 12 months
  A composite rate of target-vessel myocardial infarction (TV-MI)
Number of participants with all revascularization | 12 months
  A composite rate of all revascularization
Number of participants with ischemic driven target lesion revascularization (ID-TLR) | 12 months
  A composite rate of ischemic driven target lesion revascularization (ID-TLR)
Number of participants with stent thrombosis | Within 24 hours, 30 days, 12 months
  A composite rate of stent thrombosis
Number of participants with non-ischemic targeted lesion perfusion | 12 months
  A composite rate of non-ischemic targeted lesion perfusion
Number of participants with Non target vessel myocardial infarction | 12 months
  A composite rate of Non target vessel myocardial infarction

CONTACTS AND LOCATIONS:
Overall Officials: Deok-Kyu Cho, MD, PhD, Principal Investigator — Yongin Severance Hopistal
Locations (1):
- Yongin Severance Hospital, Yongin, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No
The data set is available from the the corresponding author upon reasonable request.